CLINICAL TRIAL: NCT02255201
Title: A Randomized, Double-Blind, Crossover Clinical Trial Comparing the Effects of Four Pre-Workout Beverages on Muscular Strength and Endurance and Cognitive Performance in Healthy Adult Males
Brief Title: Pre-Workout on Exercise Performance and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miami Research Associates (Network)
Collaborators: Glanbia Performance Nutrition (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: GPN-2014
Record Dates: First submitted 2014-09-26; First posted 2014-10-02 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- Beverage A (Active Comparator): Single dose, Pre-Workout Master Performance Blend Dose 1
  Interventions: Dietary Supplement: Master Performance Blend Dose 1
- Beverage B (Active Comparator): Single dose, Pre-Workout Master Performance Blend Dose 2
  Interventions: Dietary Supplement: Master Performance Blend Dose 2
- Beverage C (Active Comparator): Single dose, Pre-Workout Performance Energy Blend
  Interventions: Dietary Supplement: Performance Energy Blend
- Beverage D (Active Comparator): Single dose, Pre-Workout Energy Blend
  Interventions: Dietary Supplement: Energy Blend
- Beverage E (Placebo Comparator): Single dose, Pre-Workout Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Master Performance Blend Dose 1 — Caffeine content: 200 mg
  Arms: Beverage A
Dietary Supplement: Master Performance Blend Dose 2 — Caffeine content: 400 mg
  Arms: Beverage B
Dietary Supplement: Performance Energy Blend — Caffeine content: 175 mg
  Arms: Beverage C
Dietary Supplement: Energy Blend — Caffeine content: 200 mg
  Arms: Beverage D
Dietary Supplement: Placebo — Caffeine content: 0 mg
  Arms: Beverage E

SUMMARY:
The purpose of this study is to determine the effects of four different pre-workout beverages as compared to placebo on muscular strength and endurance, perceived energy and cognitive performance in healthy adult males.

ELIGIBILITY:
Inclusion Criteria:

1. Males, aged 18 to 40 years
2. Subject has a waist circumference ≤ 97 cm.
3. Subject is a non-smoker.
4. Subject is in good health and appropriate for exercise as determined by physical examination, medical history and ECG.
5. Subject is weight training for the 6 months prior to starting the trial.
6. Subject agrees to not use any new vitamins and/or minerals until after study completion and to not take any vitamins and/or minerals 24 hours prior to the test visits.
7. Subject agrees to not use any dietary or herbal supplements until after study completion. A 7-day washout is allowed for study inclusion.
8. Subject is willing and able to comply with the protocol including:

   * Attending 5 visits each of which is approximately 4 hours long;
   * Refraining from caffeine, over-the-counter medications and alcohol for the 24 hours prior to the test visits;
   * Refraining from weight training for the 48 hours prior and refraining from any exercise other than weight training for 24 hours prior to the test visits;
   * Refraining from taking any dietary or herbal supplements throughout the study.
9. Subject is able to understand and sign the informed consent to participate in the study.

Exclusion Criteria:

1. Subject has any of the following medical conditions:

   * active heart disease
   * uncontrolled high blood pressure (≥ 140/90 mmHg)
   * renal or hepatic impairment/disease
   * Type I or II diabetes
   * bipolar disorder
   * pulmonary disease (including current asthma)
   * Parkinson's disease
   * Seizure disorder
   * unstable thyroid disease
   * immune disorder (such as HIV/AIDS)
   * active psychiatric disorders (including anxiety disorders)
   * bleeding disorders
   * gastrointestinal ulcer disease
   * any medical condition deemed exclusionary by the Principal Investigator (PI)
2. Subject has any orthopedic problem(s) or history of musculoskeletal injury(ies) which make(s) resistance weight training contraindicated.
3. Subject has a history of cancer (except localized skin cancer without metastases) within 5 years prior to screening.
4. No prescription or chronic medication use allowed without PI discretion.
5. Subject is currently taking and unwilling to refrain from taking any over-the-counter stimulant medications/supplements (see section 2.6.2); seven-day washout required for study inclusion.
6. Subject is currently taking and unwilling to refrain from taking any over-the-counter allergy or asthma medication containing pseudoephedrine or ephedrine (see section 2.6.2); seven-day washout required for study inclusion.
7. Subject has an allergy to milk and phenylalanine, or any of the ingredients in the test product (see section 3.2.1).
8. Subject reports sensitivity to caffeine and/or beta-alanine.
9. Subject reports being a regular caffeine consumer defined as consuming > 600 mg of caffeine per day.
10. Subject exhibits evidence of hepatic or renal dysfunction as evidenced by ALT, AST, AP being ≥ two times the upper limit of normal or serum creatinine value ≥ 2.0 mg/dl or other clinically significant abnormal clinical laboratory value per PI discretion.
11. Subject has a clinically relevant abnormality as defined by the PI or interpreting physician with respect to the ECG.
12. Subject has a QTcB interval > 450 msec.
13. Subject has a history of drug or alcohol abuse in the past 12 months.
14. Subject has any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the subject or the quality of the study data.
15. Subject has taken an investigational product within 30 days of the first exercise test visit (visit 2).

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in Muscular Strength and Endurance compared to Placebo | One day
  Muscular Strength and Endurance will be measured by Bench Press and Leg Press 1-RM and repetitions to exhaustion.

SECONDARY OUTCOMES:
Change from Baseline in Cognitive Performance | Baseline to one-hour post dose and immediately post exercise
  Cognitive performance will be measured by the automated trail maker tests A and B.

OTHER OUTCOMES:
Change from Baseline in Perceived Energy and Fatigue | Baseline to one-hour post dose and immediately post exercise
  Perceived Energy and Fatigue will be measured by the Profile of Mood States.

CONTACTS AND LOCATIONS:
Locations (1):
- Miami Research Associates, Miami, Florida, United States